CLINICAL TRIAL: NCT02882425
Title: Single-center, Open-label, Phase 1 Study Consisting of a Single-dose Pilot Phase and a Randomized, Two-way Crossover, Single-dose Main Phase to Investigate the Absolute Bioavailability of a Single Oral Dose of Selexipag in Healthy Male Subjects
Brief Title: Absolute Bioavailability of a Single Oral Dose of Selexipag in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-065-110
Record Dates: First submitted 2016-08-18; First posted 2016-08-29 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects
Keywords: selexipag; bioavailability
MeSH Terms: interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intravenous selexipag (Pilot phase) (Experimental): Subjects received a 20-minute intravenous (i.v.) infusion of 50 µg selexipag
  Interventions: Drug: Selexipag for intravenous use
- Sequence A-B (Main phase) (Experimental): Subjects received a 80-minute i.v. infusion of 200 µg selexipag during Period 1, and 2 tablets of oral selexipag (total dose of 400 µg) as a single administration during Period 2. A washout period of 7 to 10 days separated the i.v. infusion from the oral administration.
  Interventions: Drug: Selexipag for intravenous use; Drug: Selexipag for oral use
- Sequence B-A (Main phase) (Experimental): Subjects received 2 tablets of oral selexipag (total dose of 400 µg) as a single administration during Period 1, and a 80-minute i.v. infusion of 200 µg selexipag during Period 2. A washout period of 7 to 10 days separated the oral administration from the i.v. infusion.
  Interventions: Drug: Selexipag for intravenous use; Drug: Selexipag for oral use

INTERVENTIONS:
Drug: Selexipag for intravenous use — Selexipag was reconstituted in sterile 0.9% w/v NaCl before infusion via an infusion pump at a rate of 2.5 µg/min.
  Other Names: ACT-293987
Drug: Selexipag for oral use — Tablet containing 200 µg of selexipag
  Other Names: ACT-293987
  Arms: Sequence A-B (Main phase); Sequence B-A (Main phase)

SUMMARY:
The primary purpose of this phase 1 study is to investigate the absolute bio-availability of a single oral dose of selexipag, i.e., to assess the amount of selexipag which reaches the blood when administered as an oral tablet (ACT-293987) compared to an intravenous administration in healthy subjects.

DETAILED DESCRIPTION:
A pilot phase was conducted in 3 male subjects before the main phase for assessment of absolute bio-availability conducted in 16 other male subjects. The pilot phase aimed to determine the intravenous dose to be used in the main phase based on safety data and pharmacokinetics data.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Aged from 18 to 45 (inclusive) at screening
* Body mass index (BMI) from 18.0 to 28.0 kg/m2 (inclusive) at screening
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests

Exclusion Criteria:

* Any contraindication to the study drug formulations
* History or presence of any disease or condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study drugs
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (F) of selexipag | From pre-dose to 72 hours post-dose
  F was calculated using the areas under the plasma concentrations curves extrapolated to infinity [AUC(0-inf)] after oral (po) and intravenous (iv) doses, obtained during the main phase, and using the following formula: AUC(0-inf)po * iv dose / AUC(0-inf)iv * oral dose
Area under the plasma concentration-time curve from time 0 to infinity [AUC(0-inf)] of selexipag | From pre-dose to 72 hours post-dose
  AUC(0-inf) was calculated from the concentration-time profile of selexipag after both oral and intravenous administration during the main phase

SECONDARY OUTCOMES:
Areas under the plasma concentration-time curve from time 0 to time t [AUC(0-t)] of selexipag and its active metabolite | From pre-dose to 72 hours post-dose
  AUC from time 0 to time t of the last measured concentration above the limit of quantification [AUC(0-t)] were calculated for selexipag and its active metabolite, from their respective concentration-time profiles, after both intravenous (pilot phase and main phase) and oral administration (main phase) of selexipag
Maximum plasma concentration (Cmax) of selexipag and its active metabolite | From pre-dose to 72 hours post-dose
  Cmax of selexipag and its active metabolite were directly obtained from the plasma concentration-time curves after both intravenous (pilot phase and main phase) and oral administration (main phase) of selexipag
time to reach maximum plasma concentration (tmax) of selexipag and its active metabolite | From pre-dose to 72 hours post-dose
  tmax of selexipag and its active metabolite were directly obtained from the plasma concentration-time curves after both intravenous (pilot phase and main phase) and oral administration (main phase) of selexipag
Terminal half-life [t(1/2)] of selexipag and its active metabolite | From pre-dose to 72 hours post-dose
  t(1/2) of selexipag and its active metabolite were calculated after both intravenous (pilot phase and main phase) and oral administration (main phase) of selexipag from the concentration-time profiles
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Priska Kaufmann, PhD, Study Director — Actelion

REFERENCES:
- [Result] Kaufmann P, Hurst N, Astruc B, Dingemanse J. Absolute oral bioavailability of selexipag, a novel oral prostacyclin IP receptor agonist. Eur J Clin Pharmacol. 2017 Feb;73(2):151-156. doi: 10.1007/s00228-016-2164-4. Epub 2016 Nov 24. PMID 27885399